CLINICAL TRIAL: NCT01050803
Title: Effectiveness of the Farsi Diabetes Self-management Education Program for People With Type 2 Diabetes: Randomized Controlled Trial
Brief Title: Effectiveness of the Farsi Diabetes Self-management Education (FDSME) Program for People With Type 2 Diabetes
Acronym: FDSME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FDSME
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Intervention studies; Program effectiveness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FDSME group (Experimental): In the FDSME group, sessions will be held interactive; and reflection in between sessions will be encouraged. Group-based problem-solving exercises will be used during the sessions. Participants receive feedback from peers and healthcare professionals at the following sessions.
  Interventions: Behavioral: FDSME group
- Control group (Active Comparator)
  Interventions: Behavioral: FDSME

INTERVENTIONS:
Behavioral: FDSME group — In the intervention group, diabetes education sessions which are designed based on the "Intervention Mapping" will be interactive and reflection in between sessions will be encouraged. Group-based problem-solving exercises will be used during the sessions. Participants receive feedback from peers and healthcare professionals at the following sessions.
  Arms: FDSME group
Behavioral: FDSME — In the intervention group, sessions which are designed based on the "Intervention Mapping" will be interactive and reflection in between sessions will be encouraged. Group-based problem-solving exercises will be used during the sessions. Participants receive feedback from peers and healthcare professionals at the following sessions.
  Arms: Control group

SUMMARY:
To evaluate the effectiveness of the Farsi diabetes self-management education program on psychosocial, lifestyle, and clinical measures in people with newly diagnosed people with type 2 diabetes and those with already-diagnosed type two diabetes who had received little self-management education. The development of the program was guided by an innovative process of intervention planning: Intervention Mapping.

DETAILED DESCRIPTION:
For designing the management program, we will use Intervention Mapping (IM) framework for systematically developing the theory and evidence based program.

Based on IM approach, this study will have seven phases:

Step 1: needs assessment (Development the problem analysis: health, quality of life, behavior, environment).

Step 2: We will develop proximal program objectives with a multidisciplinary expert panel of participants.

Step 3: After identification of the proximal program objectives, the next step will be to select theoretical methods and practical strategies based on evidence for alternative methods.

Step 4: The forth step of the program development will comprise of composing program materials and pre-testing these materials with a sample of patients at a diabetic outpatient clinic.

Step 5: By involving the future program facilitators (health care workers at outpatient clinics) a linkage system will be foreseen.

Step 6: planning for evaluation Step 7: Randomized Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes (according to the WHO criteria)
* Older than 18 years

Exclusion Criteria:

* Pregnancy
* Unable to participate in a group program (for example, housebound or unable to communicate in Farsi)
* Having reduced cognitive ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
HbA1c | within 2 years
BMI | 2 years

SECONDARY OUTCOMES:
Audit of Diabetes-Dependent Quality of Life (ADDQOL) | two years